CLINICAL TRIAL: NCT00531323
Title: Evaluation of the Pharmacokinetics and Safety of TMC125 Administered Once and Twice-Daily and Following a 2-Week-Treatment Period With Efavirenz in Male and Female Healthy Volunteers.
Brief Title: TMC 125 Blood Levels Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SSAT 024
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Pharmacokinetic; TMC125; Healthy volunteers; Efavarinz
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Group 1 (n =12): subjects will receive TMC125 400 mg once daily for 14 days followed by 14 days of washout followed by efavirenz 600 mg once daily for 14 days followed by 14 days of TMC125 400 mg once daily
  Interventions: Drug: TMC125 once daily
- 2 (Other): Group 2 (n = 12): TMC125 200 mg twice daily for 14 days followed by 14 days of washout followed by efavirenz 600 mg once daily for 14 days followed by 14 days of TMC125 200 mg twice daily
  Interventions: Drug: TMC125 twice daily

INTERVENTIONS:
Drug: TMC125 once daily — Group 1 (n =12): subjects will receive TMC125 400 mg once daily for 14 days followed by 14 days of washout followed by efavirenz 600 mg once daily for 14 days followed by 14 days of TMC125 400 mg once daily
  Arms: 1
Drug: TMC125 twice daily — Group 2 (n = 12): TMC125 200 mg twice daily for 14 days followed by 14 days of washout followed by efavirenz 600 mg once daily for 14 days followed by 14 days of TMC125 200 mg twice daily
  Arms: 2

SUMMARY:
The purpose of the study is to look at whether changing directly from one medication for HIV (efavirenz) to a new medication for HIV (TMC125) has any effect on the levels of TMC125 in the blood, compared to when TMC125 is taken without efavirenz having been taken immediately beforehand.

The study aims to help the investigators understand whether it is safe to change directly from efavirenz to TMC125 (with no gap between the treatments) in patients who need these treatments.

The study will investigate the blood levels of TMC125 when it is taken both once and twice a day.

DETAILED DESCRIPTION:
Pharmacokinetic parameters of TMC125 will be evaluated when TMC125 is given without and with a 14-day efavirenz intake preceding period in order to evaluate the risk of achieving sub therapeutic concentrations of TMC125 when switching straight from efavirenz containing regimens

Safety and tolerability of medications will also be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the drug study.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month after the study

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B and/or C antibodies
4. Positive blood screen for HIV-1 and 2 antibodies
5. Current or recent (within 3 months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
7. Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug
8. Consumption of grapefruit, or Seville oranges or any grapefruit or Seville orange containing product within 1 week of first dose of study drug and for the duration of the study
9. Use of any other drugs, including over-the-counter medications and herbal preparations, within 2 weeks prior to first dose of study drug
10. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period
11. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of TMC125 administered once and twice-daily and following a 2-week-treatment period with efavirenz 600 mg once daily | 56 days

SECONDARY OUTCOMES:
Efavirenz inducing effect on TMC125 metabolism after efavirenz intake cessation evaluation. Safety and tolerability of TMC125 administered once and twice-daily | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — Chelsea & Westminser Healthcare NHS Trust
Locations (1):
- St Stephens Centre, Chelsea & Westminster Hospital, London, United Kingdom